CLINICAL TRIAL: NCT05230823
Title: Acceptability of the Small Changes Behavioural Weight Loss Approach for Patients with Atrial Fibrillation and Obesity in Cardiac Rehabilitation
Brief Title: Behavioural Weight Loss Treatment for Patients with Atrial Fibrillation and Obesity in Cardiac Rehabilitation
Acronym: BE-WEL in CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-1437
Record Dates: First submitted 2021-11-23; First posted 2022-02-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation; Obesity
MeSH Terms: conditions — Atrial Fibrillation; Obesity

STUDY DESIGN:
Intervention Model Description: This novel intervention will be tested in a single group study using a pre-post intervention design prior to testing in a large RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The intervention consists of a traditional 12-week outpatient CR program with added weekly behavioural weight loss classes.
  Interventions: Behavioral: CR with added BWLT

INTERVENTIONS:
Behavioral: CR with added BWLT — 12 week outpatient cardiac rehab (CR) program consisting of twice-weekly supervised exercise and risk factor modification (e.g. smoking cessation, support with medication). Concurrently, the patients will attend a weekly behavioural weight loss treatment (BWLT). Weekly goal-setting facilitated by the interventionist will focus on behavioural changes in nutrition and moderate calorie reduction while also emphasizing physical activity consistent with an individualized CR exercise prescription. Patients will track caloric intake, weekly exercise, weekly weight, and success/challenges with other health goals (e.g., challenging negative thoughts, body image, mindful eating, etc.) using a daily health diary. ASPIRE-AF will be delivered virtually to small groups (8-12 patients) by senior PhD students with advanced training in cognitive-behavioural therapy and motivational communication principles.

SUMMARY:
One-in-four Canadians will be diagnosed with an abnormal heart rhythm called atrial fibrillation (AF) in their lifetime. People with AF have an increased chance of having serious medical problems like stroke and heart failure. Nearly three-quarters of people with AF also have obesity (excess body weight). According to research, people with obesity that lose approximately 10% of their body weight can experience relief from uncomfortable AF symptoms. Losing weight may even help people return to a normal heart rhythm.

Cardiac rehabilitation (CR) is a proven way to help people with heart disease live longer, healthier lives. So far, research has not shown whether CR helps improve the abnormal heart rhythms seen in AF. This may be because CR programs usually do not offer specific help with weight management. Therefore, adding behavioural weight-loss treatment (BWLT; group classes to change thoughts and behaviours to encourage weight-loss) to CR programs may help people with AF and obesity experience relief from their symptoms.

This study will test a new BWLT provided within a traditional CR program. Patients who have AF and obesity will take traditional CR with added BWLT. Traditional CR consists of participating in exercise sessions, supervised by health professionals, twice per week for 12 weeks. In addition to exercising, patients will complete 12 online group therapy classes to learn strategies from psychology to help them lose weight. After patients complete the 12 week program the investigators will collect patients' perspectives on the program in order to make changes if needed before testing BWLT in a larger group of people. The investigators will also weigh patients and measure their AF symptoms before and after the program to determine if taking CR+BWLT helps with weight loss and AF symptoms. This research will help efforts to provide effective treatment to patients with AF to help them lose weight and reduce or eliminate AF symptoms.

DETAILED DESCRIPTION:
Background: One-in-four Canadians will develop atrial fibrillation (AF), increasing risk of heart failure and stroke. Obesity (i.e., BMI ≥30 kg/m2) represents a strong, independent risk factor for increased incidence and severity of AF. Weight loss reduces AF symptom burden, and patients with obesity who lose ≥10% of their body weight may achieve AF regression/remission. Cardiac rehabilitation (CR) improves AF risk factors including hypertension and cardiorespiratory fitness (CRF), yet the efficacy of CR for reducing AF symptom burden is not established. CR rarely includes targeted obesity management and, on average, has a negligible impact on BMI. Adding behavioural weight-loss treatment (BWLT) to traditional CR may therefore enhance weight loss and lead to improvements in AF prognosis, symptoms, and health-related quality-of-life (HRQOL) in patients with AF and obesity.

A recent qualitative investigation of potential barriers and facilitators to patient uptake of a BWLT+CR intervention demonstrated that a combined CR+BWLT program is desirable to patients with AF and obesity. Results of this study will be used to adapt the existing small changes BWLT to meet the unique needs of this patient population prior to testing the intervention. Demonstrating that an AF adapted-version of the BWLT, delivered during a traditional 12-week CR program, is acceptable to patients with AF and comorbid obesity is a necessary next-step in intervention development, prior to testing the intervention in randomized designs.

The primary aim is to: Demonstrate acceptability of an adapted 12-week BWLT program, provided in the context of 12-weeks of exercise-based CR, among patients with AF and obesity.

The secondary aims of the proposed study are to: (a) Evaluate the feasibility of the fixed BWLT protocol in terms of recruitment, retention, drop out rates, treatment protocol adherence (by interventionists), and intervention adherence (attendance at BWLT and CR completion), and (b) evaluate potential improvements in weight, AF symptom burden, and psychological distress (depression, anxiety) from pre- to post-BWLT+CR program.

Hypotheses:

The primary study hypothesis is that patients will find the AF-adapted BWLT+CR program acceptable, as evidenced by ≥80% satisfaction with the intervention on the post-intervention assessments.

Secondary hypotheses are that: patients will demonstrate reductions in weight, BMI, waist circumference (when measured), AF symptom burden, as well as improved psychological distress from pre- to post- intervention.

Study design:

Design and Procedure. Patients will be assessed for eligibility at the Calgary AF clinic and TotalCardiology Rehabilitation (TCR). Eligible patients who consent to participate will be enrolled into the CR program and scheduled for the next available BWLT group session. Prior to their first BWLT session, patients will complete a questionnaire battery including socio-demographic variables (age, sex, ethnicity, income, education), self-reported weight and height to establish BMI, and validated questionnaires assessing AF symptom burden, AF-related quality-of-life, general HRQOL, and psychological distress at baseline (T1). Patients will be re-administered the test battery following the 12-week BWLT program (T2). (Note: T2 measures will be administered even if the patient is still completing their remaining CR exercise sessions. CR completion/adherence will be determined after patients have completed their 12-week exercise program). Additionally, intervention acceptability will be assessed using a patient survey at T2. Weight loss from baseline to 12-weeks will be calculated and converted to a percentage of initial body weight at baseline. Clinical variables (e.g., CRF from graded exercise tests; blood pressure, lipids) will be obtained by TCR chart review.

Recruitment. Patients will be recruited in three ways: (1) directly from the Calgary AF clinic using referrals from co-investigator S. Wilton, (2) from TotalCardiology Rehabilitation, and (3) from an existing database of patients who participated in the Part I qualitative study who provided consent to be contacted about future studies. The recruitment period will be November 2021 to May 2022. Equal numbers of men and women will be recruited. AF clinic patients who are both (a) eligible for the CR program and (b) eligible for the propose study will be identified by Dr. Wilton and/or AF clinic staff. Dr. Wilton/AF clinic staff will inform patients who meet (a) and (b) criteria about the study and invite them to participate. Interested patients will receive a CR referral and their contact information will be provided to the research coordinator. The research coordinator (T. Williamson) will contact patients, provide additional information about the study, and obtain informed consent. The research coordinator will then schedule patients for the next available BWLT session and send an email link to complete baseline questionnaires. Concurrently, patients will be contacted by CR staff to schedule their orientation appointment, as per typical clinic procedures. This recruitment procedure will also apply to patients who previously participated in Part I (i.e the qualitative study).TCR patients who are currently enrolled in CR will also be recruited. A research team member will identify CR patients who have consented to be approached about research and who are eligible for inclusion by reviewing patient chart data. An RA will contact patients by telephone to review study procedures and obtain patients' informed consent. Patients who agree to participate will be scheduled for the next available BWLT session and e-mailed a link to complete the study questionnaire battery (T1) online via Qualtrics Software system. Patients will be instructed to complete the questionnaire battery prior to attending the first BWLT session.

Sample Size/Analysis. Analysis will be by intention to treat. Powering early-phase studies to detect statistically significant effects is not typically recommended. A final sample of 30 (15 women) will be used; 40 patients will be recruited to allow for a 25% LTFU. The primary outcome of intervention acceptability will be evaluated using descriptive statistics of acceptability survey responses and qualitative analysis of patients' open-field responses. Feasibility outcomes will also be assessed through descriptive statistics reporting adherence, drop out, recruitment, and fidelity rates. The secondary outcome of weight change will be evaluated in a within-subjects mixed (Gender; Time) ANOVA. Changes in additional secondary and exploratory variables will be evaluated in within-subjects mixed ANOVAs.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years
* symptomatic, electrocardiogram (ECG)-documented paroxysmal (i.e., ≥2 AF episodes within a 6 month period) or persistent (i.e., AF episodes lasting ≥7 days) AF
* obesity (i.e., BMI ≥30 kg/m2)
* able to read and write in English to be eligible.

Exclusion Criteria:

* longstanding-persistent (i.e., ≥ 3 years continuous AF) or permanent AF;
* uncontrolled CAD;
* currently enrolled in a concurrent weight loss program, and;
* currently scheduled to receive catheter ablation treatment for AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability | Post-intervention (12 weeks)
  Patients will be surveyed to asses satisfaction with the intervention
Intervention Feasibility | Post-intervention (12 weeks)
  Adherence to the intervention will be determined by chart review. Referral rates of eligible patients from the AF clinic will be recorded. Drop-outs will be recorded, including reasons for study drop-out if available. The clinical supervisor (Dr. Rouleau) will evaluate the interventionists' adherence to the BWLT manual and provide feedback as needed (e.g., regarding adherence to the manual, therapeutic/process skills).

SECONDARY OUTCOMES:
Weight Loss | baseline, 12-weeks
  Patients will be weighed before and after the 12 week intervention and weight loss calculated in kilograms
Atrial Fibrillation Symptom Burden | Baseline, 12-weeks
  University of Toronto AF Symptoms Severity Scale (AFSS) - The AFSS assesses subjective and objective AF disease burden across four domains: AF burden (frequency, duration, and severity of AF episodes); global well being (visual analogue scale where patients rate their life from "worst" to "best" 1-10)
AF-related quality of life | baseline, 12-weeks
  Atrial Fibrillation Effect on Quality-of-Life Questionnaire (AFEQT) - The AFEQT is a 20-item self-report questionnaire assessing impact of AF across four QOL domains: symptoms, daily activities, treatment concern, and treatment satisfaction. A large (6-centre) prospective validation study indicates the AFEQT has high (> 0.88) internal consistency, and is sensitive to intervention effects (i.e., scores increased 3-month post-ablation). Lower AFEQT scores are associated with increased AF severity.
Symptoms of Psychological Distress | baseline, 12-weeks
  Symptoms of depression will be measured using the Beck Depression Inventory-II (BDI-II) a 21-item self-report questionnaire with well-established cut-offs for minimal, mild, moderate, and severe depressive symptoms. Symptoms of anxiety will be measured using the Beck Anxiety Inventory (BAI), a 21-item self-report scale assessing severity of anxious symptoms over the past month on a 0-3 point Likert scale. The BAI has good reliability (i.e., one-week test-retest reliability = 0.75 and Cronbach's α = 0.92) and established cut-offs for low, moderate, and high anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Tavis S Campbell, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No